CLINICAL TRIAL: NCT02006719
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of AA4500 for the Treatment of Adhesive Capsulitis of the Shoulder
Brief Title: Clinical Study for the Treatment of Adhesive Capsulitis of the Shoulder
Acronym: AC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUX-CC-871
Record Dates: First submitted 2013-12-02; First posted 2013-12-10 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
Keywords: Adhesive Capsulitis; Frozen Shoulder; Shoulder Range of Motion limitation; Shoulder Pain
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase Clostridium Histolyticum (Experimental): Up to 3 injections of .58 mg/1 mL of collagenase clostridium histolyticum (CCH), minimum of 21 days apart and home shoulder exercise.
  Interventions: Biological: Collagenase Clostridium Histolyticum
- Placebo (Placebo Comparator): Up to 3 1-mL injections of placebo, minimum of 21 days apart and home shoulder exercise.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Collagenase Clostridium Histolyticum — Treatment of Adhesive Capsulitis
  Other Names: AA4500; Xiaflex; Xiapex
  Arms: Collagenase Clostridium Histolyticum
Other: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the safety, effectiveness, and immunogenicity of AA4500 in the treatment of adhesive capsulitis.

DETAILED DESCRIPTION:
Study is a Phase 2b, double-blind, placebo-controlled study of the safety and efficacy of AA4500 for the treatment of adhesive capsulitis of the shoulder. To be eligible for treatment, a subject must have unilateral idiopathic adhesive capsulitis of the shoulder with restricted range of motion in the affected shoulder for at least 3 months but not more than 12 months. Subjects will be screened for study eligibility within 28 days before injection of study drug.

Approximately 300 adult women and men are to be enrolled in this study. Following screening and determination of study eligibility, subjects will be randomized 3:1 to receive 0.58 mg of AA4500 or placebo. Subjects will receive up to 3 injections of study drug. Each injection will be separated by a minimum of 21 days. Subjects will also be instructed in home shoulder exercises after the first injection.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral idiopathic adhesive capsulitis of one shoulder for at least 3 months but not more than 12 months (Frozen Stage)
* Normal range of motion in the contralateral shoulder
* Restricted active range of motion (AROM) in the affected shoulder defined as: a deficit of at least 60 degrees in total AROM in the affected shoulder as compared with the total AROM in the contralateral shoulder and a deficit of at least 30 degrees in AROM in at least one of the following planes as compared with the contralateral shoulder:

  * Forward flexion
  * Abduction
  * External rotation with the elbow up to 90 degrees abduction
  * Internal rotation with the elbow up to 90 degrees abduction

Exclusion Criteria:

* Has received treatment for adhesive capsulitis or is planning to receive treatment for adhesive capsulitis at any time during the study including but not limited to:

  * physical therapy or acupuncture within 2 weeks before the first injection of study drug
  * intra-articular or intrabursal injection(s) of lidocaine; suprascapular nerve blocks; corticosteroids, electroanalgesic and/or thermoanalgesic modalities within 1 month before the screening visit
  * intra-articular or intrabursal injection(s) of sodium hyaluronate and/or glenohumeral distension arthrography within 3 months before the screening visit
  * surgical intervention (including shoulder manipulation under anesthesia) at any time
* Has any of the following conditions, as determined by investigator to be potentially confounding to the evaluation of safety and efficacy:

  * Adhesive capsulitis as a result of traumatic injury (ie, direct injury to the shoulder such as fracture of the humerus or clavicle immediately preceding the onset of this episode of adhesive capsulitis). Traumatic events in the past that are not temporally related to the onset of this episode of adhesive capsulitis would not necessarily exclude a subject from participating in the study.
  * Active subacromial impingement in the affected shoulder
  * Calcified tendonitis in the affected shoulder
  * Glenohumeral joint arthritis in the affected shoulder
  * Arthrosis of the affected shoulder
  * Chondrolysis of the affected shoulder
  * Subscapularis tendon rupture of the affected shoulder
  * Other rotator cuff injuries of the affected shoulder
  * Uncontrolled hypertension
  * Uncontrolled diabetes
  * Uncontrolled thyroid disease
  * History of thrombosis or post-thrombosis syndrome
  * Physical impairment that would preclude performing the protocol defined exercises
  * Active infection in area to be treated
  * Clinically significant neurological disease
  * Bleeding disorder
  * Chronic use of anticoagulation medications and the subject cannot be cleared medically to stop taking medication for 7 days prior to each injection. Less than or equal to 150 mg aspirin is allowed during the study.
  * Known active hepatitis A, B, or C
  * Other significant medical condition (eg, morbid obesity, cervical disc disease), which in the investigator's opinion would make the subject unsuitable for enrollment in the study
* Has received oral or intravenous steroids for any reason within 3 weeks before the screening visit
* Has received an investigational drug or treatment within 30 days before the first dose of study drug.
* Has a known allergy to collagenase or any other excipient of AA4500 or any other procedural medication.
* Has, at any time, received collagenase for the treatment of adhesive capsulitis.
* Is unable to undergo an x-ray or MRI (contraindication) evaluation of the affected shoulder.
* Is planning to be treated with commercial XIAFLEX at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil H Schusterman, MD FACP, Study Director — Endo Pharmaceuticals
Locations (46):
- United States (35):
  - Alabama Orthopaedic Center-Research, Birmingham, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Advance Med Clinical Research, Carlsbad, California
  - Triwest Research Associates, El Cajon, California
  - Core Orthopedic Medical Center, Encinitas, California
  - Temecula Rheumatology & Internal Medicine, Murrieta, California
  - Clearview Medical Research, Santa Clarita, California
  - Colorado Orthopedic Consultants, PC, Englewood, Colorado
  - Florida Research Associates, DeLand, Florida
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - Jewett Orthopedic Clinic, Orlando, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Non-Surgical Orthopedics, P.C. / Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Injury Care Medical Center, Boise, Idaho
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Rockford Orthopedics Associates, Rockford, Illinois
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - PRN of Kansas, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Bone and Joint Clinic, Gretna, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - Arthritis and Rheumatism Associates, PC, Wheaton, Maryland
  - Great Falls Clinic, Great Falls, Montana
  - Nevada Orthopedic & Spine Center, Las Vegas, Nevada
  - Stony Brook University Medical Center (SUNY), Stony Brook, New York
  - Triangle Orthopedic Associates, PA, Durham, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - The Neuromusculoskeletal Center of the Cascades d.b.a. The Center, Bend, Oregon
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - University of Pennsylvania Penn Orthopaedics, Philadelphia, Pennsylvania
  - Texas Orthopedic Specialist, Bedford, Texas
  - Centex Studies, Houston, Texas
  - Commonwealth Orthopaedics & Rehabilitation, Arlington, Virginia
  - Danville Orthopedic Clinic, Inc., Danville, Virginia
- Australia (11):
  - Sports Medicine Professionals, Richmond, Victoria
  - Hunter Clinical Research, NSW
  - Royal Prince Alfred, NSW
  - St George Hospital, NSW
  - Peninsula Private Hospital, Queensland
  - QPharm, Queensland
  - Menzies Research Institute, Tasmania
  - Emeritus Research, VIC
  - Epworth Hospital, VIC
  - Repatriation Hospital, VIC
  - Hand and Upper Limb Centre, WA

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500: Up to 3 injections of 0.58 mg/1 mL collagenase clostridium histolyticum (AA4500), minimum of 21 days apart and home shoulder exercise
- Placebo: Up to three 1-mL injections of placebo, minimum of 21 days apart and home shoulder exercise
Period: Overall Study
Arm/Group | AA4500 | Placebo
Started | 237 | 85
Completed | 219 | 80
Not Completed | 18 | 5
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Other/Unknown | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 administration of study drug (1 participant excluded)
Groups:
- AA4500: Up to 3 injections of 0.58 mg/1 mL AA4500, minimum of 21 days apart and home shoulder exercise
- Total: Total of all reporting groups
Arm/Group | AA4500 | Placebo | Total
Number analyzed (Participants) | 237 | 84 | 321
Age, Continuous [Median (Full Range); unit: years] | 53.0 [29 to 75] | 51.0 [22 to 70] | 52.0 [22 to 75]
Age, Customized [Count of Participants; unit: Participants]
  <45 | 30 | 14 | 44
  45-54 | 114 | 44 | 158
  55-64 | 75 | 23 | 98
  65-74 | 17 | 3 | 20
  ≥75 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 60 | 222
  Male | 75 | 24 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 4 | 21
  Not Hispanic or Latino | 220 | 80 | 300
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 22 | 7 | 29
  White | 205 | 72 | 277
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 95 in Active Forward Flexion
Description: Active range of motion (AROM) measurement using a goniometer to assess forward flexion in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 active forward flexion measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 41.0 (28.89) | 35.9 (23.36)

2. Secondary Outcome: Change From Baseline to Day 95 in Adapted American Shoulder and Elbow Surgeons (ASES) Function Subscale
Description: Function subscale score ranging from 0-50, with 0 being most dysfunctional, derived from participant assessment of ability to do 10 activities with affected shoulder/arm where 0=unable to do to, 1=very difficult to do, 2=somewhat difficult, and 3=not difficult, and calculated as (cumulative total score for the 10 activity items) × (5/3); adapted from ASES Standardized Shoulder Assessment Form, Patient Self-Evaluation (United States adapted version).
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 34 participants missing either baseline or day 95 function subscale scores also excluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 211 | 76
units on a scale | 17.0 (11.65) | 14.8 (11.14)

3. Secondary Outcome: Change From Baseline to Day 95 in Pain With Movement Using 11-point Numeric Rating Scale (NRS)
Description: Participant assessment of pain in response to "How bad is the pain upon movement of your affected shoulder at its worst in the last 24 hours?" using an 11-point NRS where 0=no pain at all and 10=pain as bad as it can be.
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 33 participants missing either baseline or day 95 pain with movement scores also excluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 211 | 77
units on a scale | -4.4 (2.83) | -3.9 (2.93)

4. Secondary Outcome: Change From Baseline to Day 95 in Active Abduction
Description: AROM measurement using a goniometer to assess abduction in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 active abduction measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 49.0 (33.10) | 43.8 (30.71)

5. Secondary Outcome: Change From Baseline to Day 95 in Passive Forward Flexion
Description: Passive range of motion (PROM) measurement using a goniometer to assess forward flexion in the affected shoulder
Time Frame: Baseline, day 95
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 39.3 (29.47) | 34.1 (22.37)

6. Secondary Outcome: Change From Baseline to Day 95 in Passive Abduction
Description: PROM measurement using a goniometer to assess abduction in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 passive abduction measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 45.4 (33.69) | 42.8 (32.12)

7. Secondary Outcome: Change From Baseline to Day 95 in Active Internal Rotation
Description: AROM measurement using a goniometer to assess internal rotation in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 active internal rotation measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 23.1 (25.21) | 20.9 (23.58)

8. Secondary Outcome: Change From Baseline to Day 95 in Active External Rotation
Description: AROM measurement using a goniometer to assess external rotation in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 active external rotation measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 28.6 (21.30) | 26.1 (22.67)

9. Secondary Outcome: Change From Baseline to Day 95 in Passive Internal Rotation
Description: PROM measurement using a goniometer to assess internal rotation in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 passive internal rotation measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 24.1 (23.77) | 20.3 (23.61)

10. Secondary Outcome: Change From Baseline to Day 95 in Passive External Rotation
Description: PROM measurement using a goniometer to assess external rotation in the affected shoulder
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 25 participants missing either baseline or day 95 passive external rotation measurement also excluded
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 217 | 79
degrees | 24.8 (22.31) | 24.4 (26.16)

11. Secondary Outcome: Change From Baseline to Day 95 in Adapted ASES Pain Subscale
Description: Pain subscale score ranging from 0-50, with 0 being greatest pain, derived from participant overall assessment of pain in response to "How bad is the pain in your affected shoulder today?" using an 11-point NRS where 0=no pain at all and 10=pain as bad as it can be and calculated as (10 - NRS score) x 5; adapted from ASES Standardized Shoulder Assessment Form, Patient Self-Evaluation
Time Frame: Baseline, day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 33 participants missing either baseline or day 95 pain subscale scores also excluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 211 | 77
units on a scale | 15.9 (13.46) | 13.5 (13.45)

12. Secondary Outcome: Subject Satisfaction With Treatment at Day 95
Description: Participant assessment of satisfaction with treatment rated as very satisfied, quite satisfied, neither satisfied nor dissatisfied, quite dissatisfied, or very dissatisfied.
Time Frame: Day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 11 participants not completing questionnaire also excluded
Measure: Number; unit: participants
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 229 | 81
participants
  Very satisfied | 142 | 43
  Quite satisfied | 38 | 22
  Neither satisfied nor dissatisfied | 32 | 8
  Quite dissatisfied | 10 | 2
  Very dissatisfied | 7 | 6

13. Secondary Outcome: Investigator Assessment of Improvement With Treatment at Day 95
Description: Investigator assessment of degree of improvement in severity of the participant's treated shoulder compared with screening rated as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Time Frame: Day 95
Population: All participants who have a baseline AROM measurement of the affected shoulder and at least 1 measurement of AROM of the affected shoulder following the first administration of study drug (1 participant excluded); 10 participants also excluded for incomplete questionnaire
Measure: Number; unit: participants
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 229 | 82
participants
  Very much improved | 94 | 27
  Much improved | 73 | 31
  Minimally improved | 41 | 16
  No change | 13 | 8
  Minimally worse | 6 | 0
  Much worse | 1 | 0
  Very much worse | 1 | 0

ADVERSE EVENTS:
Time Frame: 130 days (up to 28 day screening period and 95±7 day study period)
Arm/Group | AA4500 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/237 | 1/84
Other Adverse Events (participants affected / at risk) | 188/237 | 37/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=237) | Placebo (N=84)
Atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=237) | Placebo (N=84)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 90 (138) | 18 (24)
Contusion (Injury, poisoning and procedural complications) | 71 (106) | 2 (2)
Injection site bruising (General disorders) | 52 (65) | 10 (13)
Injection site pain (General disorders) | 50 (77) | 11 (17)
Ecchymosis (Skin and subcutaneous tissue disorders) | 47 (69) | 3 (4)
Localised oedema (General disorders) | 20 (28) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (16) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes